CLINICAL TRIAL: NCT03031067
Title: Comparison Between Hypothermic Oxygenated Perfusion and Static Cold Storage of Organ From Extended Criteria Donors
Brief Title: Hypothermic Oxygenated Perfusion Versus Static Cold Storage for Marginal Graft
Acronym: PIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matteo Ravaioli (Other)
Responsible Party: Sponsor-Investigator, Matteo Ravaioli, Principal Investigator, University of Bologna
Organization: University of Bologna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIO-700; 159/2015/O/Disp (Registry Identifier: ID ethics committee)
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Liver Diseases; Kidney Diseases
Keywords: Donors and donation; Extended criteria donor; Organ perfusion and preservation; Liver transplantation; Kidney transplantation; Preservation injury; Ischemia reperfusion injury
MeSH Terms: conditions — Liver Diseases; Kidney Diseases; Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: A matched-case analysis was developed: 10 HOPE-ECD livers and kidneys, HOPE-L and -K groups, were matched 1:3 with livers and kidneys preserved with static cold storage (SCS), SCS-L and -K groups respectively.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Machine perfusion - Kidney (Experimental): The marginal kidney will be perfused with oxygenated solution of preservation at 4°C for two hours with Exiper, Bologna Machine Perfusion.
  Interventions: Device: Machine perfusion
- Static cold storage - Kidney (No Intervention): The marginal kidney that was stored to cold (SCS), previously.
- Machine perfusion - Liver (Experimental): The marginal liver will be perfused with oxygenated solution of preservation at 4°C for two hours with Exiper, Bologna Machine Perfusion.
  Interventions: Device: Machine perfusion
- Static cold storage - Liver (No Intervention): The marginal liver that was stored to cold (SCS), previously.

INTERVENTIONS:
Device: Machine perfusion — The graft preservation will be performed perfusing with a oxygenated solution of preservation at 4°C for two hours with Exiper, Bologna Machine Perfusion, developed by Medica s.p.a and our research group.
  Flow and pressure values will be set up for the kidney and liver perfusion, differently. The oxygenation of solution will be performed by an oxygenator and a filter for decapneization / oxygenation. During the perfusion the oxygen pressure will be required between 600-750 mmHg (pO2 80-100 Kpa), as reported in the scientific literature. The pH, lactate concentration, and oxygen (PO2) and carbon dioxide (PCO2) partial pressure were measured in the preservation solution at T0 and T1 by means of a standard haemogasanalyzer.
  Other Names: Hypothermic Oxygenated Perfusion
  Arms: Machine perfusion - Kidney; Machine perfusion - Liver

SUMMARY:
One of the major challenge in the field of organ transplantation is the shortage of donor organs. Many patients waiting for organ transplantation die during the waiting time and many patients wait for organ transplantation many years with a detrimental effect on their quality of life, and increasing morbidity and the costs related to. Effective strategies, which safely extends the donor pool, are therefore advocated. During the last 20 years the two main policies to gain this purpose were the living donation and the utilization of extended donor's criteria (ECD). These donors are supposed to yield a lower outcome than the conventional donors and many research protocols were developed to reduce the preservation injury (PI) and PI-related complications. Static cold storage (SCS) has been the standard technique in clinical practice for liver and kidney preservation using particular solutions (Wisconsin, Custodiol and Celsior) able to prevent cellular swelling. Recently, graft preservation with hypothermic machine perfusion (HMP) is developing, because it seems to improve early graft function due to increased tissue ATP concentrations upon reperfusion and due to the continual flush of the microcirculation which removes waste products.

The addition of oxygen during the perfusion represents an innovation in the methods of preservation in approved clinical setting seems to add further improvements of the graft. The present study was designed in order to assess the impact of hypothermic oxygenated perfusion (PIO) of marginal human kidney and liver compared with SCS.

DETAILED DESCRIPTION:
Our national single-center study, interventional with medical device, exploratory and safety, will be assessed the optimal graft preservation, liver and kidney, from marginal donors ECD (Expanded Criteria Donors), using hypothermic oxygenated perfusion (PIO) compared to the static cold storage that is the preservation control method of custom. PIO will be applied to 10 ECD liver transplants and 10 ECD kidney transplants that meet the inclusion criteria.

The marginal graft will be perfused with oxygenated solution of preservation at 4°C for two hours with Exiper, Bologna Machine Perfusion, developed by Medica s.p.a and our research group.

Flow and pressure values will be set up for the kidney and liver perfusion, otherwise. The oxygenation of solution will be performed by an oxygenator and a filter for decapneization / oxygenation. During the perfusion the oxygen pressure will be required between 600-750 mmHg (pO2 80-100 Kpa), as reported in the scientific literature. The pH, lactate concentration, and oxygen (PO2) and carbon dioxide (PCO2) partial pressure were measured in the preservation solution at T0 and T1 by means of a standard haemogasanalyzer.

After transplantation, the recipients will be monitored clinically to assess the graft function. The liver's data will be compared with similar case treated with SCS in our centre of transplant, retrospectively; instead, the kidney's data will be compared with the "twin" organ transplanted without PIO, prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Kidney donor: ECD.
* Kidney recipient: single or dual kidney transplant recipients at our center, provided consent.
* Liver donor: ECD
* Liver recipient: liver transplant recipients at our center, provided consent.

Exclusion Criteria:

* Kidney donor: no ECD, donor with vascular anatomical abnormalities and/or urinary tract, donor with a risk infection, to increase cold ischemia time can not be avoided.
* Kidney recipient: patients with severe atherosclerotic vascular disease, pathologies predisposing to the onset of intra-operative surgical complications, such as thrombophilia and hemophilia, antigenic incompatibility with donor determining the acute rejection of the organ; patients waiting for kidney transplant pre-emptive, multi-organ transplant, retransplantation.
* Liver donor: no ECD, donor with vascular anatomical abnormalities, donor with a risk infection, to increase cold ischemia time can not be avoided.
* Liver recipient: patients with acute liver disease and with vascular abnormalities and/or biliary tract requiring non-conventional reconstructive techniques, patients waiting for multi-organ transplant, retransplantation, urgency transplant ( or with MELD>30).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Graft function | 3 months post-transplantation (+18/-2 months)
  Physiological values of serum creatinine and diuresis for kidney transplantation and bilirubin, AST, ALT, INR for liver transplantation

SECONDARY OUTCOMES:
Graft survival - Kidney | 3 months post-transplantation (+18/-2 months)
  Time (days) of graft survival
Graft survival - Liver | 3 months post-transplantation (+18/-2 months)
  Time (days) of graft survival
Patient survival (kidney recipient) | 3 months post-transplantation (+18/-2 months)
  Time (days) of patient survival
Patient survival (liver recipient) | 3 months post-transplantation (+18/-2 months)
  Time (days) of patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Ravaioli, PhD, Principal Investigator — University of Bologna S. Orsola-Malpighi Hospital, Transplantation and General Surgery Unit; Antonio Daniele Pinna, Professor, Study Director — University of Bologna S. Orsola-Malpighi Hospital, Transplantation and General Surgery Unit
Locations (1):
- Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be performed by application of a single code.

REFERENCES:
- [Background] O'Callaghan JM, Morgan RD, Knight SR, Morris PJ. Systematic review and meta-analysis of hypothermic machine perfusion versus static cold storage of kidney allografts on transplant outcomes. Br J Surg. 2013 Jul;100(8):991-1001. doi: 10.1002/bjs.9169. PMID 23754643
- [Background] Thuillier R, Allain G, Celhay O, Hebrard W, Barrou B, Badet L, Leuvenink H, Hauet T. Benefits of active oxygenation during hypothermic machine perfusion of kidneys in a preclinical model of deceased after cardiac death donors. J Surg Res. 2013 Oct;184(2):1174-81. doi: 10.1016/j.jss.2013.04.071. Epub 2013 May 21. PMID 23731682
- [Background] Hosgood SA, Nicholson HF, Nicholson ML. Oxygenated kidney preservation techniques. Transplantation. 2012 Mar 15;93(5):455-9. doi: 10.1097/TP.0b013e3182412b34. PMID 22217529
- [Background] Dutkowski P, Polak WG, Muiesan P, Schlegel A, Verhoeven CJ, Scalera I, DeOliveira ML, Kron P, Clavien PA. First Comparison of Hypothermic Oxygenated PErfusion Versus Static Cold Storage of Human Donation After Cardiac Death Liver Transplants: An International-matched Case Analysis. Ann Surg. 2015 Nov;262(5):764-70; discussion 770-1. doi: 10.1097/SLA.0000000000001473. PMID 26583664